CLINICAL TRIAL: NCT04318509
Title: Market Research - Acceptability Study for a New PKU Glycomacropeptide Based Protein Substitute (Dr Schär- Mevalia Amino Acids) Mevalia PKU GMPower - Vanilla
Brief Title: Market Research - Acceptability Study for a New PKU Protein Substitute
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Schär AG / SPA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GMPower1
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: PKU; Phenylketonurias; Inborn Errors of Metabolism; Metabolic Disease
MeSH Terms: conditions — Phenylketonurias; Metabolism, Inborn Errors; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PKU GMPOWER (Experimental): (casein) glycomacropeptide protein substitute for the dietary management of PKU from the age of 3 years
  Interventions: Dietary Supplement: GMPOWER

INTERVENTIONS:
Dietary Supplement: GMPOWER — (casein) glycomacropeptide protein substitute for the dietary management of PKU from the age of 3 years

SUMMARY:
The aim of this study is to demonstrate that a new protein substitute is acceptable and well tolerated in children with PKU.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PKU or PKU variant requiring a protein substitute.
* Subjects who were already taking a phenylalanine-free/low phenylalanine protein substitute and were willing to try the study product for 7 days.
* Patients aged 3 years of age to adulthood.
* Written informed consent obtained from participant or parental caregiver (as appropriate).

Exclusion Criteria:

* Presence of serious concurrent illness
* Investigator's uncertainty about the willingness or ability of the patient to comply with the protocol requirements
* Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.
* Any patients having taken antibiotics over the previous 2 weeks leading up to the study.
* Patients less than 3 years of age.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-05-19 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | 7 days
  Questionnaire detailing any GI symptoms, severity and change from usual
  • The collection of daily data about the gastro-intestinal tolerance of the protein substitute.
Product compliance | 7 days
  Daily questionnaire on amounts offered and amounts actually consumed, compared to recommended amount.
Product palatability | 7 days
  Questionnaire data captured to evaluate taste
Product acceptability | 7 days
  Brief tick-box questionnaire on overall liking and acceptability of product

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol

IPD SHARING:
Plan to Share IPD: No